CLINICAL TRIAL: NCT06385392
Title: Continuous Wearable Monitor for the Detection and Release of Freezing of Gait.
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Other Study IDs: A23-354
Record Dates: First submitted 2024-04-22; First posted 2024-04-26 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
Keywords: Freezing of Gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with Parkinson's disease and Freezing of Gait using experimental insole and haptic module
  Interventions: Device: Haptic module and insole device

INTERVENTIONS:
Device: Haptic module and insole device — System for use in daily in-community use that detects the occurrence of freezing of gait (FOG) and triggers external cueing stimuli to unfreeze the individual.

SUMMARY:
The proposed system (haptic module and insole device) for daily in-community use that detects the occurrence of freezing of gait (FOG) in people with Parkinson's disease (PD). and triggers external cueing stimuli to unfreeze the individual. The purpose of the overall Phase II study is to: (1) Develop a production ready system, (2) Develop a companion mobile app for the proposed system and refine previously developed FOG detection algorithms, and (3) Validate the proper operation of the system and demonstrate its efficacy through lab and in-community testing. This study will focus on validating the system and demonstrating efficacy through in-community testing.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide and provision of signed and dated informed consent form.
* Age 45 or older
* Diagnosis of idiopathic PD, as determined by a movement disorders neurologist in accordance with the PD Society Brain Bank diagnostic criteria.
* Evidence of presence of freezing gait as a symptom. Determined from combination of clinical examination (observation of freezing) and New Freezing of Gait Questionnaire (NFOG).
* Able to complete a 2-minute walk test at the pre-treatment visit.
* Currently on a stable prescription medication regimen for PD and willing to adhere to the regimen during the study.
* Ability to don and doff the insole and haptic module independently or have daily assistance during the study intervention.

Exclusion Criteria:

* Non-English speaking
* History of musculoskeletal disorders that significantly affect movement of lower limbs as determined at the time of enrollment.
* Other significant neurological disorders that may affect participation or performance in the study.
* Neuropathy at the ankle assessed at the pre-treatment visit using the haptic module.
* Hallucinations
* Non-ambulatory
* Legally Blind
* Symptomatic hypotension
* Any condition which would limit sensation in the legs or requires use of wraps, bandages or other items which may limit sensation in the legs (e.g., lymphedema) that would interfere with the performance of the haptic device, in the opinion of the investigator.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants aged 45-80 who have a diagnosis of Parkinson's disease with Freezing of Gait symptoms who live in the community.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
To validate the haptic module and insole device system and evaluate its efficacy with an in-community clinical trial. | 5 weeks
  Change in duration of FOG events. Decreased duration of FOG events indicates higher efficacy of device system.

CONTACTS AND LOCATIONS:
Overall Officials: Martha A Nance, MD, Principal Investigator — Struthers Parkinson's Center
Locations (2):
- United States (2):
  - Struthers Parkinson's Center, Golden Valley, Minnesota
  - HealthPartners Neuroscience Center, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No